CLINICAL TRIAL: NCT01804998
Title: Multicenter Phase III Trial of Laparoscopic Sentinel Node Biopsy and Stomach Preserving Surgery in Early Gastric Cancer
Brief Title: Multicenter Phase III Trial of Laparoscopic Sentinel Node Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Keun Won Ryu, Principal investigator, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SENORITA 2013
Record Dates: First submitted 2013-03-04; First posted 2013-03-05 (Estimated); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Early Gastric Cancer
Keywords: laparoscopic sentinel lymph node biopsy; phase 3; early gastric cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: Stomach preserving surgery after laparoscopic sentinel node dissection and evaluation
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic Sentinel Node Biopsy (Experimental): Laparoscopic Sentinel Node Biopsy or Stomach Preserving Surgery could be performed in this arm
  Interventions: Procedure: Laparoscopic Sentinel Node Biopsy
- Laparoscopy Assisted Gastrectomy (Active Comparator): Conventional procedure is laparoscopy assisted gastrectomy in early gastric cancer patient.
  Interventions: Procedure: Laparoscopy Assisted Gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic Sentinel Node Biopsy — Laparoscopic Sentinel Node Biopsy or Stomach Preserving Surgery could be performed in the experimental arm.
  Arms: Laparoscopic Sentinel Node Biopsy
Procedure: Laparoscopy Assisted Gastrectomy — In the control arm, laparoscopy assisted gastrectomy with lymph node dissection (D1+ or more) will be performed.
  Arms: Laparoscopy Assisted Gastrectomy

SUMMARY:
Laparoscopic sentinel lymph node biopsy and stomach preserving surgery in early gastric cancer is less invasive method which can increase quality of life. For last two years, multicenter quality control study (Phase II) has been performed in Korea and tolerable results were observed. Based on these results, multicenter phase III trial is required to validate the clinical role of laparoscopic sentinel lymph node biopsy.

DETAILED DESCRIPTION:
The final analyses include the modified intention to treatment analysis (full analysis set) and Per Protocol analysis (including patients who underwent assigned surgery without agreement withdrawal).

1. Injection of tracer and sentinel basin dissection

   * Tracer: Tc 99m HSA (Human serum albumin, 2ml, 0.1mCi/ml) + ICG (indocyanine green, 2ml, 5mg/ml)
   * Endoscopic injection of tracer on 4 sites around gastric cancer
   * Identification of sentinel basin using laparoscopic probe (Neoprobe)
   * Laparoscopic sentinel basin dissection and identification of sentinel node at back table
2. Surgical considerations

   * If positive sentinel nodes were diagnosed in frozen section, conventional gastrectomy is performed.
   * If micrometastasis or isolate tumor cells in sentinel basin lymph nodes were diagnosed in the permanent pathology, re-operation of conventional gastrectomy is not performed.
   * However, re-operation of converntional gastrectomy should be performed in case of macrometastasis, deep and lateral margin positive, more than pT2 lesion in the permanent pathology.
3. H.pylori eradication - There was no clear evidence that H.pylori eradication reduced development of metachronous gastric cancer. H.pylori eradication was planned to perform according to physician's decision or patient's need. However, recently, the effect of H.pylori eradication in development of metachronous gastric cancer was published in NEJM (Choi et al. 2018). Therefore, from now on, H. pylori eradication will be recommended to enrolled patients with H.pylori.

ELIGIBILITY:
Inclusion Criteria:

* single lesion of adenocarcinoma in preoperative endoscopic biopsy
* clinical stage T1N0 in the preoperative evaluation of endoscopy and computed tomography
* tumor size: less than 3cm
* location: 2cm far from the pylorus or cardia
* aged 20 to 80
* ECOG 0 or 1
* patient who signed the agreement
* patient who is suspected to underwent laparoscopy assisted gastrectomy

Exclusion Criteria:

* indication of endoscopic submucosal resection
* inoperable due to poor cardiac, pulmonary function
* pregnant
* having allergic reaction, previous upper abdominal surgery except laparoscopic cholecystectomy, previous radiation therapy to upper abdomen
* diagnosed as malignancy within 5 years except carcinoma in situ of cervix cancer and thyroid cancer

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 580 (Actual)
Dates: Start 2013-03-27 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
3 year disease free survival rate | 3 years after surgery
  A total of enrollment period is suspected to be four years and patients will be followed up for five years. However, primary end point is 3 year disease free survival and we can analyze survival data at three year later from when the last enrolled patients underwent intervention.

SECONDARY OUTCOMES:
postoperative morbidity and mortality | 30 days after surgery
  We will collect morbidity and mortality data for postoperative 30 days. Therefore, this end point will be completed one month later from when the last enrolled patients underwent intervention.
scores of global health status scale, functional scales, and symptom scales/items of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ) C30 and STO22 | 3 years
  Survey for quality of life will be performed regularly for three years after surgery. Measurement tool is the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ) C30 and STO22. In EORTC QLQ C30, there are 1 global health status scale, 5 functonal scales, and 9 symptom scales/items. EORTC QLQ STO22 includes 5 symptom scales and 4 single items. Each scale and item ranges 0 to 100. Higher score of global health status and functinoal scales indicate better quality of life and lower score of symptom scales indicates better quality of life. There is no summed score in these questionnaires.
5 year disease free survival rate | 5 years after surgery
  A total of enrollment period is suspected to be four years and patients will be followed up for five years. Therefore, we can complete data collection at five year later from when the last enrolled patients underwent intervention
5 year overall survival rate | 5 years after surgery
  A total of enrollment period is suspected to be four years and patients will be followed up for five years. Therefore, we can complete data collection at five year later from when the last enrolled patients underwent intervention
3 year recurrence free survival rate | 3 years after surgery
  A total of enrollment period is suspected to be four years and patients will be followed up for five years. However, primary end point is 3 year disease free survival and we can analyze survival data at three year later from when the last enrolled patients underwent intervention.
3 year disease specific death rate | 3 years after surgery
  A total of enrollment period is suspected to be four years and patients will be followed up for five years. However, primary end point is 3 year disease free survival and we can analyze survival data at three year later from when the last enrolled patients underwent intervention.
3 year overall survival rate | 3 years after surgery
  3 years after surgery
5 year recurrence free survival rate | 5 years after surgery
  A total of enrollment period is suspected to be four years and patients will be followed up for five years. Therefore, we can complete data collection at five year later from when the last enrolled patients underwent intervention.
5 year disease specific death rate | 5 years after surgery
  A total of enrollment period is suspected to be four years and patients will be followed up for five years. Therefore, we can complete data collection at five year later from when the last enrolled patients underwent intervention

CONTACTS AND LOCATIONS:
Locations (7):
- South Korea (7):
  - Chonnam National University Hwasun Hospital, Hwasun, Chonnam
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Soonchunhyang University Bucheon Hospital, Bucheon-si
  - Dongnam Institute of Radiological and Medical Science, Busan
  - Gyeongsang National University, Jinju
  - Yonsei Univeristy College of Medicine, Seoul
  - Ajou University School of Medicine, Suwon

IPD SHARING:
Plan to Share IPD: Undecided
We will discuss this topic in the research meeting later.

REFERENCES:
- [Derived] Eom BW, Yoon HM, Kim YW, Min JS, An JY, Hur H, Lee YJ, Cho GS, Park YK, Jung MR, Park JH, Hyung WJ, Jeong SH, Kook MC, Han M, Nam BH, Ryu KW; Sentinel Node Oriented Tailored Approach (SENORITA) Study Group. Quality of Life and Nutritional Outcomes of Stomach-Preserving Surgery for Early Gastric Cancer: A Secondary Analysis of the SENORITA Randomized Clinical Trial. JAMA Surg. 2024 Aug 1;159(8):900-908. doi: 10.1001/jamasurg.2024.1210. PMID 38809537
- [Derived] Kim YW, Min JS, Yoon HM, An JY, Eom BW, Hur H, Lee YJ, Cho GS, Park YK, Jung MR, Park JH, Hyung WJ, Jeong SH, Kook MC, Han M, Nam BH, Ryu KW. Laparoscopic Sentinel Node Navigation Surgery for Stomach Preservation in Patients With Early Gastric Cancer: A Randomized Clinical Trial. J Clin Oncol. 2022 Jul 20;40(21):2342-2351. doi: 10.1200/JCO.21.02242. Epub 2022 Mar 24. PMID 35324317
- [Derived] An JY, Min JS, Hur H, Lee YJ, Cho GS, Park YK, Jung MR, Park JH, Hyung WJ, Jeong SH, Kim YW, Yoon HM, Eom BW, Kook MC, Han MR, Nam BH, Ryu KW; SEntinel Node ORIented Tailored Approach (SENORITA) Study Group. Laparoscopic sentinel node navigation surgery versus laparoscopic gastrectomy with lymph node dissection for early gastric cancer: short-term outcomes of a multicentre randomized controlled trial (SENORITA). Br J Surg. 2020 Oct;107(11):1429-1439. doi: 10.1002/bjs.11655. Epub 2020 Jun 3. PMID 32492186
- [Derived] Park JY, Kim YW, Ryu KW, Nam BH, Lee YJ, Jeong SH, Park JH, Hur H, Han SU, Min JS, An JY, Hyung WJ, Cho GS, Jeong GA, Jeong O, Park YK, Jung MR, Yoon HM, Eom BW. Assessment of laparoscopic stomach preserving surgery with sentinel basin dissection versus standard gastrectomy with lymphadenectomy in early gastric cancer-A multicenter randomized phase III clinical trial (SENORITA trial) protocol. BMC Cancer. 2016 May 31;16:340. doi: 10.1186/s12885-016-2336-8. PMID 27246120